CLINICAL TRIAL: NCT01133145
Title: Allogenic Vascularized Knee and Femur Transplantation Clinical Evaluation
Brief Title: Allogeneic Vascularized Knee Transplantation
Acronym: kneeTx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Jena (Other)
Responsible Party: Michael Diefenbeck, MD, clinic of trauma, hand and reconstructive surgery, University of Jena
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: knee Tx
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2010-05

CONDITIONS: Osteitis; Limb Salvage; Joint Deformities, Acquired; Skin Transplantation; Bone Transplantation
Keywords: composite tissue allotransplantation; hand transplantation; knee transplantation; face transplantation
MeSH Terms: conditions — Osteitis; Joint Deformities, Acquired

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- vascularized transplantation (Experimental): allogeneic vascularized knee transplantation
  Interventions: Procedure: knee joint transplantation

INTERVENTIONS:
Procedure: knee joint transplantation — transplantation of a kne joint from a multi organ donor to a recipient with a severly injured knee joint

SUMMARY:
High energy trauma often results in severe soft tissue, bone and joint injury. Today, many methods and techniques exist to treat theses severely injured extremities. Surgical techniques include open reduction and internal fixation (ORIF), e.g. with screws and plates, soft tissue reconstruction by local or free flaps and joint reconstruction by arthroplasty, e.g. total knee arthroplasty. In few, very severe cases, those methods are not sufficient to restore function and amputation is the only option left.

In 1908 the German surgeon Erich Lexer had the idea to transplant a joint. Due to the medical situation at his time the attempts failed.

But the idea survived and was processed over the time. Transplant surgery and medicine developed, immunosuppressive drugs were established and animal models proved that bone and joint transplantation is technically feasible.

In 1998 the first successful hand and in 2005 the first partial face transplantation was carried out. In 1996 we started our clinical femur and knee joint transplantation project.

DETAILED DESCRIPTION:
Sterile osseous defects of the knee joint are temporarily stabilised with a hinge arthroplasty or an intramedullary nail in the case of a long femoral defect.

Assisted passive motion and isometric exercises are possible and necessary to avoid contractions and muscular atrophy during waiting time. Informed consent has to be obtained.

The knee joint is harvested in accordance with standard organ procurement guidelines used in multi-organ donation (MOD). Authorization for knee donation must be obtained from the donor's families. MODs older than 45 years or those who had an accident involving the same leg are excluded. For additional safety reasons, MODs who had received blood substitutes or fresh-frozen plasma are excluded as well.

Harvesting of the knee joint includes perfusion of the External Iliac Artery with 4 L University of Wisconsin (UW) solution at 4°C, dissection of the femoral artery and vein distally to the proximal level of the adductor canal, transsection of the muscles and osteotomy of the femur, tibia and fibula.

To restore normal appearance of the donor leg a polyethylene spacer is inserted into the bone defect and the skin closed.

The graft then is stored in sterile conditions in three layers of plastic bags at 4° C in UW-solution.

Allograft preparation involves dissection from the surrounding soft tissue with the quadriceps tendon and the articular capsule intact, vessels perfusing the muscles ligated and vessels to the bone preserved.

The graft arterial pedicle is perfused with methylene blue to confirm adequate perfusion for transplantation.

The surgical procedure commences with removal of the spacer or nail. The graft is inserted and fixed by an anterograde femoral and a retrograde tibial interlocking compression nail.

The grafts vessels are anastomosed to the recipient's superficial femoral artery and vein using the end-to-side technique. Reperfusion commences immediately while the ligaments and tendons (Quadriceps Tendon, Iliotibial Tract, Gastrocnemius, Hamstrings) were reconstructed.

Immunosuppression is started immediately after reperfusion of the graft and consists of Antithymocyte Globulin (ATG), 4mg / kg bw i.v. as an induction, FK 506 (Tacrolimus; 10mg p.o.), Mycophenolate Mofetil (MMF; 2g p. o.)and Methylprednisolone, 250mg i.v. for the first 3 days. Oral Double-Drug maintenance therapy is continued with MMF (2g p.o.) and FK 506 (Tacrolimus) with a serum level between 8 and 10 µg/ml from the beginning of the third week.

ELIGIBILITY:
Inclusion Criteria:

* severly injured knee joint with the combination of: massive bone defect plus articulating cartilage defect plus insufficient extensor mechanism (injury of patella, patella ligament or quadriceps tendon)

Exclusion Criteria:

* active osteomyelitis
* history of malignoma
* contraindications for immunosuppressive medication

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Primary Completion 2011-12 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
survival of graft | 2 years after transplantation
  Clinical examination of graft, x-rays

CONTACTS AND LOCATIONS:
Overall Officials: Gunther O Hofmann, Prof. Dr., Study Director — Clinic of Trauma-, Hand, and Reconstructive Surgery, University of jena
Locations (1):
- Klinik für Unfall-, Hand- und Wiederherstellungschirurgie, Universitätsklinikum Jena, Jena, Germany

REFERENCES:
- [Result] Hofmann GO, Kirschner MH, Wagner FD, Brauns L, Gonschorek O, Buhren V. Allogeneic vascularized transplantation of human femoral diaphyses and total knee joints--first clinical experiences. Transplant Proc. 1998 Sep;30(6):2754-61. doi: 10.1016/s0041-1345(98)00803-3. PMID 9745561
- [Result] Hofmann GO, Kirschner MH. Clinical experience in allogeneic vascularized bone and joint allografting. Microsurgery. 2000;20(8):375-83. doi: 10.1002/1098-2752(2000)20:83.0.co;2-0. PMID 11150987
- [Result] Kirschner MH, Brauns L, Gonschorek O, Buhren V, Hofmann GO. Vascularised knee joint transplantation in man: the first two years experience. Eur J Surg. 2000 Apr;166(4):320-7. doi: 10.1080/110241500750009186. PMID 10817331
- [Result] Hofmann GO, Kirschner MH, Brauns L, Wagner FD, Land W, Buhren V. Vascularized knee joint transplantation in man: a report on the first cases. Transpl Int. 1998;11 Suppl 1:S487-90. doi: 10.1007/s001470050525. PMID 9665043
- See also: University of Jena, Medicine — http://www.uniklinikum-jena.de